CLINICAL TRIAL: NCT00386308
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multicenter Study To Evaluate Efficacy and Safety of XP12B for the Treatment of Menorrhagia
Brief Title: Efficacy and Safety Study of XP12B in Women With Menorrhagia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP12B-MR-303
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2010-02-22 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2010-06

CONDITIONS: Menorrhagia; Heavy Menstrual Bleeding
Keywords: Heavy Menstrual Bleeding; Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Tranexamic acid tablets
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Tranexamic acid tablets — 3900 mg/Day
  Other Names: Lysteda; XP12B
  Arms: 1
Drug: Placebo tablets
  Other Names: Lysteda; XP12B
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether XP12B is effective and safe in the treatment of women with heavy menstrual bleeding associated with menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* Women with menorrhagia
* 18-49 years of age
* Regularly occurring menstrual periods

Exclusion Criteria:

* History or presence of clinically significant disease or abnormalities that may confound the study
* History of bilateral oophorectomy or hysterectomy
* Hormone therapy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (49):
- United States (49):
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, Carmichael, California
  - Investigative Site, San Diego, California
  - Investigative Site, Upland, California
  - Investigative Site, Denver, Colorado
  - Investigative Site, Lakewood, Colorado
  - Investigative Site, Groton, Connecticut
  - Investigative Site, West Hartford, Connecticut
  - Investigative Site, Inverness, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Decatur, Georgia
  - Investigative Site, Savannah, Georgia
  - Investigative Site, Idaho Falls, Idaho
  - Investigative Site, Amite, Louisiana
  - Investigative Site, Baton Rouge, Louisiana
  - Investigative Site, Marrero, Louisiana
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Paw Paw, Michigan
  - Investigative Site, Scottsbluff, Nebraska
  - Investigative Site, Lawrenceville, New Jersey
  - Investigative Site, Canfield, Ohio
  - Investigative Site, Centerville, Ohio
  - Investigative Site, Cleveland, Ohio
  - Investigative Site, Zanesville, Ohio
  - Investigative Site, Norman, Oklahoma
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Eugene, Oregon
  - Investigative Site, Medford, Oregon
  - Investigative Site, Portland, Oregon
  - Investigative Site, Salem, Oregon
  - Investigative Site, Abington, Pennsylvania
  - Investigative Site, Jenkintown, Pennsylvania
  - Investigative Site, Reading, Pennsylvania
  - Investigative Site, Charleston, South Carolina
  - Investigative Site, Columbia, South Carolina
  - Investigative Site, Greenville, South Carolina
  - Investigative Site, Greer, South Carolina
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Knoxville, Tennessee
  - Investigative Site, Memphis, Tennessee
  - Investigative Site, Dallas, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Sandy City, Utah
  - Investigative Site, Spokane, Washington
  - Investigative Site, Charleston, West Virginia
  - Investigative Site, Huntington, West Virginia
  - Investigative Site, Menomonee Falls, Wisconsin

REFERENCES:
- [Derived] Bushnell DM, Martin ML, Moore KA, Richter HE, Rubin A, Patrick DL. Menorrhagia Impact Questionnaire: assessing the influence of heavy menstrual bleeding on quality of life. Curr Med Res Opin. 2010 Dec;26(12):2745-55. doi: 10.1185/03007995.2010.532200. Epub 2010 Nov 3. PMID 21043553
- [Derived] Lukes AS, Moore KA, Muse KN, Gersten JK, Hecht BR, Edlund M, Richter HE, Eder SE, Attia GR, Patrick DL, Rubin A, Shangold GA. Tranexamic acid treatment for heavy menstrual bleeding: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):865-875. doi: 10.1097/AOG.0b013e3181f20177. PMID 20859150

RESULTS

PARTICIPANT FLOW:
Groups:
- 3900 mg/Day: Two 650 mg Lysteda (tranexamic acid) tablets taken 3 times daily (3900 mg/day) for a maximum of 5 days during monthly menstruation
- Placebo: Two placebo tablets taken 3 times daily for a maximum of 5 days during monthly menstruation
Period: Overall Study
Arm/Group | 3900 mg/Day | Placebo
Started | 123 | 73
Intent to Treat Population | 117 | 72
Modified Intent to Treat Population | 115 | 72
Completed | 94 | 54
Not Completed | 29 | 19
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 2 | 5
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 10 | 6
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Other Event | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3900 mg/Day | Placebo | Total
Number analyzed (Participants) | 117 | 72 | 189
Age Continuous [Mean (Standard Deviation); unit: years] — Intent to Treat Population
  years | 39 (6) | 39 (7) | 39 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 72 | 189
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Patient Reported Outcome Measure of Limitations in Social or Leisure Activities Associated With Heavy Menstrual Bleeding
Description: A positive unit change mean relects an improvement from baseline. Patient reported outcome scores had the following response categories: 1=not limited at all; 2=slightly limited; 3=moderately limited; 4=quite a bit limited; and 5=extremely limited
Time Frame: Change from Baseline scores over 6 menstrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 115 | 72
units on a scale | 0.9 (0.8) | 0.4 (0.4)

2. Secondary Outcome: Patient Reported Outcome Measure of Limitations in Physical Activities Associated With Heavy Menstrual Bleeding
Description: as for outcome 1
Time Frame: Change from Baseline scores over 6 menstrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 115 | 72
units on a scale | 0.9 (0.9) | 0.4 (0.9)

3. Secondary Outcome: Responder Analysis - Reduction in Large Stains
Description: Percentage of subjects who experienced a reduction from baseline in the frequency of large stains
Time Frame: Reduction from Baseline over 6 menstrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Number; unit: percentage of subjects
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 115 | 72
percentage of subjects | 57 | 51

4. Primary Outcome: Mean Reduction From Baseline in Menstrual Blood Loss (MBL)
Description: reduction of menstrual blood loss in mL
Time Frame: Baseline MBL over 6 menstrual cycles
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 115 | 72
mL | 66 (64) | 18 (36)

ADVERSE EVENTS:
Arm/Group | 3900 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 2/117 | 3/72
Other Adverse Events (participants affected / at risk) | 111/117 | 66/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3900 mg/Day (N=117) | Placebo (N=72)
Acute Bronchitis (Infections and infestations) | 0 | 1
Decreased Blood Sugar (Investigations) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3900 mg/Day (N=117) | Placebo (N=72)
Abdominal Pain (Gastrointestinal disorders) | 23 | 10
Anemia (Blood and lymphatic system disorders) | 12 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 28 | 14
Fatigue (General disorders) | 8 | 3
Headache (Nervous system disorders) | 69 | 39
Migraine (Nervous system disorders) | 7 | 4
Muscle Cramps & Spasms (Musculoskeletal and connective tissue disorders) | 9 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 2
Nasal & Sinus Symptoms (Respiratory, thoracic and mediastinal disorders) | 43 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other